CLINICAL TRIAL: NCT04288206
Title: Supracondylar Pinning Antibiotic Stewardship (SPAS) Trial
Acronym: SPAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Justin Brohard, Co-Investigator, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPAS Trial
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Supracondylar Humerus Fracture; Infection
Keywords: antibiotic stewardship; post operative infection; pediatric; cefazolin
MeSH Terms: conditions — Infections | interventions — Cefazolin; Saline Solution

STUDY DESIGN:
Intervention Model Description: intervention arm of intravenous cefazolin at the time of surgery (standard of care) vs placebo arm of intravenous normal saline at the time of surgery
Who Masked: Participant, Care Provider, Investigator
Masking Description: 'study drug' will be prepared by a participating pharmacist and labeled with a study identification number. The drug will be otherwise not labeled with regard to the arm of the study. This will be delivered to the operating room and administered to the patient. The patient will be entered into a spreadsheet with the study identification number to be used later to evaluate the data. The enrolling/consenting surgeon, and the patient and consenting family member, will be masked to the arm of the study throughout.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo control (Placebo Comparator): Patient will receive 'study drug' which is comprised of 300 mL of normal saline without any medication/antibiotic, which will be delivered by intravenous means at the time of surgery.
  Interventions: Drug: normal saline
- Cefazolin prophylaxis (Active Comparator): Patient will receive 'study drug' which is comprised of weight-based dose of cefazolin mixed in 300 mL of normal saline, which will be delivered by intravenous means at the time of surgery.
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — intravenous cefazolin is being evaluated as a pre-operative prophylactic antibiotic measure with primary outcome being post operative infection rate among participants.
  Arms: Cefazolin prophylaxis
Drug: normal saline — intravenous normal saline placebo
  Arms: Placebo control

SUMMARY:
Prospective, multi-center, randomized controlled trial studying infection rate with or without prophylactic antibiotics at the time of closed reduction and percutaneous pinning of pediatric supracondylar humerus fractures.

DETAILED DESCRIPTION:
The goal of the SPAS trial will be to determine the role of prophylactic antibiotics in closed reduction and percutaneous fixation of pediatric supracondylar humerus fractures. The study will be designed as a prospective, double-blinded, two-arm, non-inferiority trial. The control arm will receive standard of care preoperative prophylactic antibiotics. The intervention group will receive a preoperative saline placebo. The primary outcome of the study will be the development of a surgical site infection, including all infections both superficial and deep. Secondary outcomes will include rate and type of post-operative complications in either group, to account for any drug-related adverse outcomes. The hypothesis is that this surgery is safe to perform without prophylactic antibiotics, and the investigators anticipate finding no difference in infection rates between the two groups. Inclusion criteria will consist of an isolated, closed, displaced supracondylar humerus fracture treated with closed reduction and temporary percutaneous pinning. Immunocompromised patients, pathological fractures, open fractures, polytrauma, skeletally mature patients, and those treated primarily with open reduction or those converted to open reduction will be excluded. Because of the low infection rate observed in this type of surgery, the sample size for the study is estimated at 600 patients per arm for adequate power. With a multicenter design, the expectation will be enrollment over the course of 1-2 years with a follow up of approximately 3 months post-surgical intervention per participant.

ELIGIBILITY:
Inclusion Criteria:

* Closed, isolated extension type supracondylar humerus fracture, Gartland type 2, 3, or 4

Exclusion Criteria:

* Inability to secure consent
* Open fractures
* Polytrauma
* Pathologic fractures
* Flexion type fracture
* Associated compartment syndrome
* Allergy to cefazolin which precludes its use
* Skeletally mature patients or patients greater than 18 years of age
* Medical comorbidities including immunocompromised state, active infection, and any associated bone, endocrine, or neoplastic conditions contributing to local or generalized abnormal bone mineralization.
* Inability to attain satisfactory reduction and fixation via closed manipulation, resulting in conversion to open reduction

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
deep post operative infection | 3 months post intervention/surgery
  rate of deep post operative infections at the surgical site, requiring treatment including possible hospital admission, intravenous antibiotics, or surgical intervention
superficial post operative infection | 3 months post intervention/surgery
  rate of superficial post operative infections at the surgical site, requiring treatment limited to oral antibiotics, local wound care, pin removal, or cast change/removal

CONTACTS AND LOCATIONS:
Overall Officials: Bob Umberhandt, MD, Principal Investigator — Physician within Legacy Health System
Locations (1):
- Legacy Emanuel Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified prior to sharing amongst participating researchers. Each participating site will maintain a spreadsheet of participants with their study identification numbers. This information will be de-identified prior to sharing with the PI and safety monitor at LHS. This will occur at a midterm assessment for safety, as well as at the completion of data collection when it is time to process and analyze the data.

REFERENCES:
- [Background] Campbell KA, Stein S, Looze C, Bosco JA. Antibiotic stewardship in orthopaedic surgery: principles and practice. J Am Acad Orthop Surg. 2014 Dec;22(12):772-81. doi: 10.5435/JAAOS-22-12-772. PMID 25425612
- [Background] Prokuski L. Prophylactic antibiotics in orthopaedic surgery. J Am Acad Orthop Surg. 2008 May;16(5):283-93. doi: 10.5435/00124635-200805000-00007. PMID 18460689
- [Background] Johnson SP, Zhong L, Chung KC, Waljee JF. Perioperative Antibiotics for Clean Hand Surgery: A National Study. J Hand Surg Am. 2018 May;43(5):407-416.e1. doi: 10.1016/j.jhsa.2017.11.018. Epub 2018 Feb 3. PMID 29398330
- [Background] Formaini N, Jacob P, Willis L, Kean JR. Evaluating the use of preoperative antibiotics in pediatric orthopaedic surgery. J Pediatr Orthop. 2012 Oct-Nov;32(7):737-40. doi: 10.1097/BPO.0b013e318269543b. PMID 22955540
- [Background] Rizvi M, Bille B, Holtom P, Schnall SB. The role of prophylactic antibiotics in elective hand surgery. J Hand Surg Am. 2008 Mar;33(3):413-20. doi: 10.1016/j.jhsa.2007.12.017. PMID 18343301
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Vaquero-Picado A, Gonzalez-Moran G, Moraleda L. Management of supracondylar fractures of the humerus in children. EFORT Open Rev. 2018 Oct 1;3(10):526-540. doi: 10.1302/2058-5241.3.170049. eCollection 2018 Oct. PMID 30662761
- [Background] Iobst CA, Spurdle C, King WF, Lopez M. Percutaneous pinning of pediatric supracondylar humerus fractures with the semisterile technique: the Miami experience. J Pediatr Orthop. 2007 Jan-Feb;27(1):17-22. doi: 10.1097/bpo.0b013e31802b68dc. PMID 17195791
- [Background] Schroeder NO, Seeley MA, Hariharan A, Farley FA, Caird MS, Li Y. Utility of Postoperative Antibiotics After Percutaneous Pinning of Pediatric Supracondylar Humerus Fractures. J Pediatr Orthop. 2017 Sep;37(6):363-367. doi: 10.1097/BPO.0000000000000685. PMID 26558958
- [Background] Bashyal RK, Chu JY, Schoenecker PL, Dobbs MB, Luhmann SJ, Gordon JE. Complications after pinning of supracondylar distal humerus fractures. J Pediatr Orthop. 2009 Oct-Nov;29(7):704-8. doi: 10.1097/BPO.0b013e3181b768ac. PMID 20104149